CLINICAL TRIAL: NCT05337202
Title: The Dutch Multicentre Study Into Opportunistically Screening Geriatric Patients for Atrial Fibrillation Using a PPG Smartphone App; the Dutch-GERAF Study
Brief Title: the Dutch-GERAF Study
Acronym: GERAF
Status: Active, not recruiting | Type: Observational
Sponsor: Dijklander Ziekenhuis (Other)
Responsible Party: Sponsor
Other Study IDs: WB 694
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation; Frailty; Major Bleed
Keywords: Atrial Fibrillation; Frailty; Major Bleed; Intra cranial Haemorrhage; Cognitive disorder; eHealth
MeSH Terms: conditions — Atrial Fibrillation; Frailty; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Full blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: HeartSDK — The photoplethysmography (PPG) application enables patients to perform a finger tip heartbeat measurement and automatic analysis

SUMMARY:
Geriatric patients are at high risk of cardiovascular complications, and for the development of atrial fibrillation. Often atrial fibrillation exists in these patients without specific symptoms, and could therefore remain unknown. Furthermore, concerns exist about the bleeding profile of anticoagulation in the very elderly or frail patients.

This study applies opportunistic screening for atrial fibrillation as advised in the latest ESC Guideline on the diagnosis and management of atrial fibrillation. Furthermore, multiple bleeding risk scores will be applies, to better assess the bleeding risk in very elderly or frail patients.

ELIGIBILITY:
Inclusion Criteria:

All newly referred patients of 65 years and older that visit geriatric outpatient services are eligible (including Fall clinic, Memory clinic, Pre-operative geriatric assessment clinic, or any other geriatric outpatient clinics that are led by a geriatrician).

Exclusion Criteria:

* The patient has a pacemaker or implantable cardioverter defibrillator.
* The patient is known with a severe dementia, MoCA ≤ 15 points.
* The patient has a severe tremor, from whatever cause, and thus is unable to use the PPG based smartphone AF detection algorithm.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All newly referred patients of 65 years and older that visit a geriatric outpatient service. These will form a cohort of very elderly individuals, with multi morbidity, polypharmacy, cognitive disorders, high frailty and high risk for falling. They can also be seen as a group at high risk of cardiovascular complication and/or the development of cognitive disorders.
Sampling Method: Non-Probability Sample
Enrollment: 1075 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Newly identified cases of atrial fibrillation | The first 6 months after recruitment for the study
  PPG or ECG detected new cases of atrial fibrillation

SECONDARY OUTCOMES:
Major bleeding | From recruitment until 3 years after the recruitment of the last participant
  Major bleeding, including intra cranial haemorrhage
Stroke | From recruitment until 3 years after the recruitment of the last participant
  Stroke
Death | From recruitment until 3 years after the recruitment of the last participant
  Death
Cognitive disorder | From recruitment until 3 years after the recruitment of the last participant
  Development of dementia, categorized by aetiology, during follow up
New Atrial Fibrillation, developed after the screening period | From recruitment until 3 years after the recruitment of the last participant
  New Atrial Fibrillation, developed after the screening period

CONTACTS AND LOCATIONS:
Overall Officials: René Jansen, PhD, Principal Investigator — Northwest Hospital
Locations (6):
- Netherlands (6):
  - Rijnstate, Arnhem, Gelderland
  - Dijklander Ziekenhuis, Hoorn, North Holland
  - Noordwest ziekenhuisgroep, Alkmaar
  - Meander Medisch Centrum, Amersfoort
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request, anonymized data could be shared after approval of all principal investigators

REFERENCES:
- [Background] Zwart LAR, Germans T, Simsek S, Ruiter JH, Jansen RWMM. Atrial fibrillation, anticoagulation and major bleeding in geriatric patients at risk of falling. OBM Geriatrics 2019, Volume 3, Issue 3, doi:10.21926/obm.geriatr.1903071
- [Background] Mol D, Riezebos RK, Marquering HA, Werner ME, Lobban TCA, de Jong JSSG, de Groot JR. Performance of an automated photoplethysmography-based artificial intelligence algorithm to detect atrial fibrillation. Cardiovasc Digit Health J. 2020 Oct 22;1(2):107-110. doi: 10.1016/j.cvdhj.2020.08.004. eCollection 2020 Sep-Oct. No abstract available. PMID 35265881
- [Result] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Result] Zwart LA, Jansen RW, Ruiter JH, Germans T, Simsek S, Hemels ME. Opportunistic screening for atrial fibrillation with a single lead device in geriatric patients. J Geriatr Cardiol. 2020 Mar;17(3):149-154. doi: 10.11909/j.issn.1671-5411.2020.03.007. PMID 32280331
- [Result] Searle SD, Mitnitski A, Gahbauer EA, Gill TM, Rockwood K. A standard procedure for creating a frailty index. BMC Geriatr. 2008 Sep 30;8:24. doi: 10.1186/1471-2318-8-24. PMID 18826625
- [Result] Rockwood K, Mitnitski A. Frailty in relation to the accumulation of deficits. J Gerontol A Biol Sci Med Sci. 2007 Jul;62(7):722-7. doi: 10.1093/gerona/62.7.722. PMID 17634318
- [Result] Moraes JL, Rocha MX, Vasconcelos GG, Vasconcelos Filho JE, de Albuquerque VHC, Alexandria AR. Advances in Photopletysmography Signal Analysis for Biomedical Applications. Sensors (Basel). 2018 Jun 9;18(6):1894. doi: 10.3390/s18061894. PMID 29890749
- [Derived] Dutch-GERAF investigators; Zwart LAR, Spruit JR, Hemels MEW, de Groot JR, Pisters R, Riezebos RK, Jansen RWMM. Design of the Dutch multicentre study on opportunistic screening of geriatric patients for atrial fibrillation using a smartphone PPG app: the Dutch-GERAF study. Neth Heart J. 2024 May;32(5):200-205. doi: 10.1007/s12471-024-01868-6. Epub 2024 Apr 15. PMID 38619715

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT05337202/Prot_SAP_000.pdf